CLINICAL TRIAL: NCT01374763
Title: A Comparison of PR Oxycodone/Naloxone and PR Oxycodone After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kati Järvelä (Other)
Responsible Party: Sponsor-Investigator, Kati Järvelä, MD, PhD, Tampere University Hospital
Organization: Tampere University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R10133M; 2010-023025-37 (EudraCT Number)
Record Dates: First submitted 2011-05-26; First posted 2011-06-16 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Postoperative Pain; Opioid Related Disorders
Keywords: Naloxone; Oxycodone; Constipation; Pain, postoperative; Physiological effects of drugs; Analgesics, Opioid
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders; Constipation | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone (Active Comparator): Drug: prolonged-release oxycodone
  Interventions: Drug: Oxycodone
- Oxycodone/naloxone (Active Comparator): Prolonged-release oxycodone/naloxone
  Interventions: Drug: Prolonged-release oxycodone/naloxone

INTERVENTIONS:
Drug: Oxycodone — Prolonged-release oxycodone 10-30 mg twice daily
  Arms: Oxycodone
Drug: Prolonged-release oxycodone/naloxone — Prolonged-release oxycodone/naloxone 10-30 mg twice daily
  Arms: Oxycodone/naloxone

SUMMARY:
The aim of the study is to describe the effects of oxycodone/naloxone combination in comparison to oxycodone for the treatment of postoperative pain in patients undergoing cardiac surgery. The hypothesis is that the duration of opioid-induced bowel dysfunction and the need of laxatives will decrease.

DETAILED DESCRIPTION:
Opioid-induced bowel dysfunction is common in cardiac surgery patients postoperatively. Opioids are needed to treat severe postoperative pain, but they have troublesome side-effects such as nausea, vomiting and bowel dysfunction. These symptoms also limit the use of gastrointestinal tract for nutrition and medication. Combined prolonged-releases oxycodone and naloxone has been shown to provide as effective analgesia as PR oxycodone. Oxycodone/naloxone has also been suggested to improve bowel function without compromising analgesic efficacy.

The aim of the study is to describe the effects of oxycodone/naloxone combination in comparison to oxycodone for the treatment of postoperative pain in patients undergoing cardiac surgery. During the first three months of the study, all cardiac surgery patients will be treated with PR oxycodone. During the second part of the study (3 months), all cardiac surgery patients will be treated with PR oxycodone/naloxone. The primary end point is the duration of opioid-induced bowel dysfunction. Need of laxatives will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult cardiac surgery patient

Exclusion Criteria:

* Preoperative continuous use of laxatives
* Known anatomic or functional gastrointestinal disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Duration of opioid-induced bowel dysfunction postoperatively | Participants will be followed for the duration of hospital stay, an expected average of 5 days

SECONDARY OUTCOMES:
Need of laxatives postoperatively | Participants will be followed for the duration of hospital stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Kati Järvelä, MD, PhD, Principal Investigator — Tampere University Hospital Heart Center
Locations (1):
- Tampere University Hospital Heart Center, Tampere, Finland